CLINICAL TRIAL: NCT03856463
Title: CAREPlan: Coaches Activating, Reaching, and Engaging Patients in End-of-Life Care Plan
Brief Title: Coaches Activating Reaching and Engaging Patients
Acronym: CAREPlan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Manali Indravadan Patel, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Stanford12
Record Dates: First submitted 2019-02-22; First posted 2019-02-27 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Cancer; End-of-Life
Keywords: end of life; quality of care; cancer care delivery
MeSH Terms: conditions — Neoplasms; Death

STUDY DESIGN:
Intervention Model Description: As part of usual care, patients with cancer are assigned to services by a lay navigator and this will be the control group.
  For patients in the intervention, they will be assigned to the usual care lay navigator but will receive services by a lay navigator who is trained to engage patients in advance care planning.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group Arm (Experimental): Patients randomized into the intervention will be assigned a lay patient navigator who will provide information regarding early advance care planning, documentation of goals of care, and coordinating home-based care. The intervention arm will also receive usual care as provided by their local oncologists.
  Interventions: Behavioral: Lay Navigator Intervention; Other: Usual Care
- Control Group Arm (Active Comparator): The control group will receive usual care as provided by their local oncologists.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Lay Navigator Intervention — Patients randomized into the intervention will be assigned a lay health worker who will contact the patient to begin the intervention. The intervention includes: education on early advance care planning and documenting goals of care.
  Other Names: Intervention Group Arm
  Arms: Intervention Group Arm
Other: Usual Care — Usual care as provided by local oncologists

SUMMARY:
The purpose of the Team Based Advance Care Planning CAREPLAN program is to understand if a trained lay navigator who engages with patients with advanced stages of cancer can help patients in advance care planning, improve patient activation, satisfaction, quality of life, and the quality of end of life cancer care while also ensuring goal concordant cancer care at the end of life.

DETAILED DESCRIPTION:
Stanford Cancer Institute plans to implement and evaluate several critical elements to be in alignment with the mission of the organization to provide high value care to their patients. The CAREPLAN (Coaches Activating, Reaching, and Engaging Patients in Their End of Life Care Plan) intervention is an innovative program aimed to strengthen provider-patient relationships and facilitate whole person care about matters important to patients diagnosed with advanced stages of cancer and important to patients' support network and family. The project is intended to help establish patients' Goals of Care Plan with appropriate documentation, develop, deploy, and evaluate a model of care for patients with cancer that is intended to improve clinical outcomes and their experiences with their cancer care. The intervention provides patients with lay navigators who assist them and their families in formulating and discussing their goals of care with their health care teams in hopes to engage in shared-decision making for goal concordant care. The goal of the project is to demonstrate that there is improved documentation of goals of care, patient experiences, patient activation, quality of life, and quality of care and communication and that the program helps to improve goal concordant care receipt at the end of life.

ELIGIBILITY:
Inclusion Criteria:

* All patients who receive care at Stanford Cancer Institute and have genitourinary cancers and have received greater than 2 prior courses of chemotherapy treatment

Exclusion Criteria:

* Patients without capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Goals of Care Documentation | 12 months after patient enrollment
  Goals of Care documentation for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment.

SECONDARY OUTCOMES:
Emergency Department Visit using chart abstraction | 12 months after patient enrollment
  Emergency Department Use for each patient will be assessed by electronic health record abstraction from time of enrollment to 12 months after patient enrollment
Hospitalization Visit using chart abstraction | 12 months after patient enrollment
  Hospitalization Visits for each patient will be assessed by electronic health record abstraction from time of enrollment to 12 months after patient enrollment
Palliative care using chart abstraction | 12 months after patient enrollment
  Palliative care use for each patient will be assessed by electronic health record abstraction from time of enrollment to 12 months after patient enrollment
Hospice using chart abstraction | 12 months after patient enrollment
  Hospice for each patient will be assessed by electronic health record abstraction from time of enrollment to 12 months after patient enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Rodriguez GM, Parikh DA, Kapphahn K, Gupta DM, Fan AC, Shah S, Srinivas S, Teuteberg W, Seevaratnam B, Asuncion K, Chien J, Moore K, Ruiz SM, Patel MI. Coaches Activating, Reaching, and Engaging Patients to Engage in Advance Care Planning: A Randomized Clinical Trial. JAMA Oncol. 2024 Jul 1;10(7):949-953. doi: 10.1001/jamaoncol.2024.1242. PMID 38780960